CLINICAL TRIAL: NCT04937504
Title: Implementing a Skills Training Evidence-Based Treatment for Posttraumatic Stress Disorder in Primary Care (I-STEP)
Brief Title: Implementing a Skills Training Evidence-Based Treatment for Posttraumatic Stress Disorder in Primary Care
Acronym: I-STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-41323; K23MH117221-03 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-24 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Mental health treatment; Primary Care; STAIR intervention; webSTAIR intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAIR-PC Group (Active Comparator): Participants in the Skills Training in Affective and Interpersonal Regulation for Primary Care (STAIR-PC) group will complete five (30 minute each) therapist-led sessions in-person or via Telehealth for up to 15 weeks.
  Interventions: Behavioral: STAIR-PC Group
- WebSTAIR Group (Experimental): Participants in the WebSTAIR group will complete 10 self-guided, web-based modules for up to 15 weeks.
  Interventions: Behavioral: WebSTAIR Group

INTERVENTIONS:
Behavioral: STAIR-PC Group — Skills Training in Affective and Interpersonal Regulation for Primary Care (STAIR-PC) is a face-to-face, individual, brief (5 session) therapy adapted from the STAIR program. STAIR-PC is an appropriate treatment for individuals who have experienced traumatic stressors, and addresses symptom targets by teaching skills to improve coping with emotions and strengthen interpersonal relationships.
  Arms: STAIR-PC Group
Behavioral: WebSTAIR Group — WebSTAIR is a web-based self-help program adapted from the STAIR program for individuals who have experienced traumatic stressors. WebSTAIR contains 10 self-guided interactive modules that teach skills to improve coping with emotions and strengthen interpersonal relationships.
  Arms: WebSTAIR Group

SUMMARY:
A majority of residents in low income communities have been exposed to a potentially traumatic event, and up to half (30-50%) of trauma-exposed residents in safety net clinical settings meet criteria for posttraumatic stress disorder (PTSD). Despite this, only 13% receive treatment. Poor access to PTSD treatment is due to a shortage of mental health specialists.

This study aims to evaluate the implementation and effectiveness of a brief, cognitive-behavioral intervention for posttraumatic stress disorder (PTSD)-Skills Training in Affective and Interpersonal Regulation (STAIR)- that will be offered in Boston Medical Center (BMC)'s primary care clinics as the new standard of care following integrated behavioral healthcare (IBH) therapist training. In response to clinician capacity concerns and the impact of the COVID-19 pandemic, we will be offering the intervention in both clinician-administered and self-paced, web-administered formats. The evidence base suggests that STAIR, delivered both synchronously (in-person/telehealth STAIR) and asynchronously (webSTAIR), is associated with significant improvements in PTSD and depression symptoms.

DETAILED DESCRIPTION:
Participants who enroll in the study will be randomized to either in-person/telehealth STAIR or webSTAIR. Those who do not enroll in the study will still be able to receive STAIR in person or via telehealth as part of usual care.

Participant data will be for 9 months. Treatment plans will continue to be determined by usual care providers, the study has no involvement in any decisions regarding care. This means that a participant's IBH therapist can continue the therapy, offer a different treatment option, or refer to other services at any time in the study and after the study is completed. At any time, patients can also choose to change their treatment plans, for example from webSTAIR to in-person/telehealth STAIR, or to another treatment option in the clinic. Access to webSTAIR will be discontinued at 9 months.

The investigators hypothesize that offering a low intensity treatment for PTSD through primary care will improve access to and engagement in care for PTSD among BMC's patient population. The feasibility of two modes of treatment delivery will be compared, while gathering further evidence of the effectiveness of the intervention in our local setting. It is also hypothesized that both formats will be effective in reducing mental health symptoms, while webSTAIR may have some advantages in regard to uptake and long-term sustainability in usual care.

ELIGIBILITY:
Inclusion Criteria:

* Client seen in integrated behavioral health in Boston Medical Center's General Internal Medicine and Family Medicine clinics.
* Able to receive therapy in English (per participant report)
* Exposure to trauma (as indicated by Life Events Checklist (LEC) for the Diagnostic and Statistical Manual of Mental Disorders (DSM) DSM-5 [LEC-5])
* Subthreshold or Full Criteria for PTSD (as indicated by the PTSD Checklist Posttraumatic Stress Disorder Checklist (PCL) for the DSM-5 [PCL-5])
* Reasonable to access to technology needed to support either condition (e.g., phone, computer, internet access).

Exclusion Criteria:

* Patient is not appropriate for outpatient level of care / standard of care provided in Integrated behavioral health (IBH) per clinician judgement
* Currently receiving cognitive behavioral therapy for PTSD elsewhere e.g., cognitive processing theory (CPT), prolonged exposure (PE), eye movement desensitization and reprocessing (EMDR).
* Patient is experiencing bereavement (death of someone close) as primary clinical concern, and is therefore not a good fit for a PTSD-specific treatment at this time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Valentine, PhD, Principal Investigator — Boston Medical Center, Psychiatry Department
Locations (1):
- Boston Medical Center Clinics, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godfrey LB, Cloitre M, Elwy AR, Fortuna LR, Fuchs C, Valentine SE. Study protocol for a hybrid 1 effectiveness-implementation trial of Brief Skills Training in Affective and Interpersonal Regulation (Brief STAIR) and web-administered STAIR (webSTAIR) for posttraumatic stress disorder in integrated primary care. Contemp Clin Trials. 2023 Aug;131:107241. doi: 10.1016/j.cct.2023.107241. Epub 2023 May 25. PMID 37244367

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | STAIR-PC Group | WebSTAIR Group
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0
Period: 15 Weeks Assessment
Arm/Group | STAIR-PC Group | WebSTAIR Group
Started | 31 | 29
Completed | 26 | 20
Not Completed | 5 | 9
Not completed — Lost to Follow-up | 5 | 9
Period: 9 Months Assessment
Arm/Group | STAIR-PC Group | WebSTAIR Group
Started | 26 | 20
Completed | 23 | 18
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STAIR-PC Group | WebSTAIR Group | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.69 (14.95) | 36.28 (10.57) | 35.97 (12.92)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 0 | 4
  Female | 25 | 27 | 52
  Queer/Non Binary/Other | 2 | 1 | 3
  Declined to answer | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 23 | 22 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 19 | 37
  White | 5 | 5 | 10
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Disorder Symptoms Measured by PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms. The PCL-5 scale ranges from Not At All (0) to Extremely (4) so the PTSD checklist total scores can range from 0 to 80, where higher scores indicate higher severity of PTSD symptoms.
Time Frame: Baseline, 15 weeks, and 9 months
Population: Refer to participant flow for numbers of participants analyzed at baseline, 15 weeks, and 9 months assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAIR-PC Group | WebSTAIR Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 61.48 (10.18) | 58.28 (10.73)
  15 weeks: number analyzed (Participants) | 26 | 20
  15 weeks | 39.12 (22.32) | 36.30 (19.91)
  9 months: number analyzed (Participants) | 23 | 18
  9 months | 28.04 (21.61) | 36.39 (18.38)

2. Primary Outcome: Feasibility Based on Retention
Description: The number of participants who completed at least 90 minutes of an intervention by 15 weeks
Time Frame: 15 weeks
Population: An intent to treat analysis was done at 15 weeks on all participants who were enrolled (ie the 31 participants in the STAIR-PC group and the 29 participants in the WebSTAIR group).
Measure: Count of Participants; unit: Participants
Arm/Group | STAIR-PC Group | WebSTAIR Group
Number analyzed (Participants) | 31 | 29
Participants | 24 | 12

3. Primary Outcome: Acceptability Measured by Client Satisfaction Questionnaire (CSQ-8)
Description: The Client Satisfaction Questionnaire (CSQ-8) is an 8-item survey to measure and assess consumer satisfaction with health and human services. Response options differ for each item, the scale ranges from very negative response (1) to a very positive response (4), and the total range for the CSQ-8 can be from 1 to 32 with higher scores indicating higher satisfaction.
Time Frame: 15 weeks, 9 months
Population: The numbers of participants analyzed for this outcome at 15 weeks and 9 months is provided in the the data table and in the participant flow.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAIR-PC Group | WebSTAIR Group
Number analyzed (Participants) | 31 | 29
score on a scale
  15 weeks: number analyzed (Participants) | 26 | 20
  15 weeks | 26.6 (3.5) | 23.7 (6.3)
  9 months: number analyzed (Participants) | 23 | 18
  9 months | 26.1 (4.0) | 23.3 (5.9)

4. Secondary Outcome: General Mental Health Functioning Measured by the Brief Symptom Inventory (BSI-18)
Description: The Brief Symptom Inventory (BSI-18) is an 18-item self-report measure to assess psychological problems. The responses for each item ranges from Not At All (0) to Extremely (4), so the toal scores can range from 0 to 72. Higher total scores indicate higher severity of psychological distress.
Time Frame: Baseline, 15 weeks, 9 months
Population: Refer to participant flow for numbers of participants analyzed at baseline, 15 weeks, and 9 months assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAIR-PC Group | WebSTAIR Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 37.77 (16.40) | 37.21 (15.00)
  15 weeks: number analyzed (Participants) | 26 | 20
  15 weeks | 25.80 (16.65) | 28.30 (14.29)
  9 months: number analyzed (Participants) | 23 | 18
  9 months | 20.13 (17.57) | 25.29 (15.76)

5. Secondary Outcome: Emotional Regulation Measured by the Difficulties in Emotion Regulation Scale (DERS)
Description: The Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-report measure of emotion regulation difficulties. Individual item responses range from Almost never (1) to Almost always (5), creating a potential total score range for the DERS of 36 to 180. Higher total scores indicate higher symptom severity.
Time Frame: Baseline, 15 weeks, 9 months
Population: Refer to participant flow for numbers of participants analyzed at baseline, 15 weeks, and 9 months assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAIR-PC Group | WebSTAIR Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 106.26 (23.47) | 109.83 (28.28)
  15 weeks: number analyzed (Participants) | 26 | 20
  15 weeks | 92.56 (28.52) | 97.80 (28.58)
  9 months: number analyzed (Participants) | 23 | 18
  9 months | 80.87 (32.80) | 87.35 (22.77)

6. Secondary Outcome: Trauma Symptoms as Assessed by the Trauma Symptoms of Discrimination Scale (TSDS) of Discrimination Scale,
Description: The TSDS assesses discriminatory distress and anxiety-related trauma symptoms. It includes 21 items, each of which is rated on a 4-point scale ranging from 1 (Never) to 4 (Often). The total score of the TSDS is calculated by adding up the scores from all items and can range from 21 to 84. HIgher scores are asociated with more trauma.
Time Frame: Baseline, 15 weeks, 9 months
Population: Refer to participant flow for numbers of participants analyzed at baseline, 15 weeks, and 9 months assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAIR-PC Group | WebSTAIR Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 58.39 (16.61) | 56.34 (16.07)
  15 weeks: number analyzed (Participants) | 26 | 20
  15 weeks | 53.08 (16.99) | 48.30 (16.57)
  9months: number analyzed (Participants) | 23 | 18
  9months | 49.83 (18.48) | 55.38 (19.17)

7. Secondary Outcome: Social Functioning Measured by the Interpersonal Support Evaluation List - 12-item Version (ISEL-12)
Description: The Interpersonal Support Evaluation List - 12-item version (ISEL-12) is a 12-item self-report measure to assess perceptions of social supports. Each item response ranges from Definitely false (1) to Definitely true (4), creating a total score range of 12 to 48. Higher total scores indicate greater social supports.
Time Frame: Baseline, 15 weeks, 9 months
Population: Refer to participant flow for numbers of participants analyzed at baseline, 15 weeks, and 9 months assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAIR-PC Group | WebSTAIR Group
Number analyzed (Participants) | 31 | 29
score on a scale
  Baseline | 30.48 (7.54) | 31.26 (7.71)
  15 weeks: number analyzed (Participants) | 26 | 20
  15 weeks | 32.36 (9.00) | 31.77 (7.74)
  9 months: number analyzed (Participants) | 23 | 18
  9 months | 34.14 (6.81) | 33.50 (9.55)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | STAIR-PC Group | WebSTAIR Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04937504/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT04937504/ICF_000.pdf